CLINICAL TRIAL: NCT00000858
Title: Detection of Human Immunodeficiency Virus Type 1 (HIV-1) in Vaginocervical Secretions: Correlation With Clinical Status, Virologic and Immunologic Parameters, and the Presence of Other Infections
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: DATRI 009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Vagina
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To correlate HIV-1 viral load in vaginocervical secretions (VCS), as measured by culture and nucleic acid detection, with that found in peripheral blood and HIV clinical status. To determine whether systemic and local HIV specific antibody influences the quality and type of virus isolated from VCS. To ascertain whether the presence of specific infectious agents (e.g., HPV, HSV, CMV, etc.) influences the amount and type of virus isolated from VCS.

Predictors for the development of the acquired immunodeficiency syndrome (AIDS) in HIV infected individuals have been studied primarily among adult males and in selected small populations. Although many of these predictors may be relevant to women, HIV infection does manifest itself differently between the sexes. Therefore, it is important to study the spectrum of HIV disease in women and to identify unique and common markers, cofactors, and predictors of disease progression.

DETAILED DESCRIPTION:
Predictors for the development of the acquired immunodeficiency syndrome (AIDS) in HIV infected individuals have been studied primarily among adult males and in selected small populations. Although many of these predictors may be relevant to women, HIV infection does manifest itself differently between the sexes. Therefore, it is important to study the spectrum of HIV disease in women and to identify unique and common markers, cofactors, and predictors of disease progression.

Part 009: HIV-infected female adults, independent of CD4+ cell count, will provide blood and VCS specimens obtained at a single study visit, regardless of ovulatory phase.

NOTE: Subjects in this study will be patients who are currently enrolled in a multisite longitudinal study, Women's Interagency HIV Study (WIHS), which is designed to elucidate the natural history of infection with HIV-1 in U.S. women. Participation in DATRI 009 will require additional blood at the patient's scheduled WIHS visit.

Part 009a: Consent will be obtained from 65 women to allow additional evaluations to be completed on their reserve VCS specimen and on an additional peripheral blood specimen, specifically obtained for DATRI 009a during their 009 visit. An additional 8 ml CPT tube will be collected from these patients, bringing their total blood volume to 32 ml at their scheduled WIHS visit.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Premenopausal status.
* Intact uterus and cervix.
* Documented HIV infection.
* Current enrollment in a multisite longitudinal study, Women's Interagency HIV Study (WIHS).

Required:

* Stable or no antiretroviral therapy within 1 month prior to study entry.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antifungal or antimicrobial medication in the vagina.

Prior Medication:

Excluded:

* Antimicrobial or antifungal medications during the 48 hours prior to study entry.
* Use of spermicide or douche in the 48 hours prior to entry.

Coital interaction during the 48 hours prior to study visit, as reported by subject and confirmed by a negative seminal fluid assay result.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350

CONTACTS AND LOCATIONS:
Overall Officials: Reichelderfer P, Study Chair; Kovacs A, Study Chair
Locations (3):
- United States (3):
  - Univ of California / San Francisco, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York